CLINICAL TRIAL: NCT02248220
Title: Observation of the Efficacy and Tolerability of Sifrol® (Pramipexole) in Patients With Advanced Idiopathic Parkinson's Disease
Brief Title: Efficacy and Tolerability of Sifrol® (Pramipexole) in Patients With Advanced Idiopathic Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 248.360
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Pramipexole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Parkinson's disease patients
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole
  Other Names: Sifrol®

SUMMARY:
Assessment of daily maintenance dose of Sifrol®, L-dopa sparing effect, effect on tremor, depression, anhedonia and tolerability

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced idiopathic Parkinson's disease for whom combined treatment with Sifrol and L-dopa was indicated

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced idiopathic Parkinson's diease recruited at specialist practices and hospitals
Sampling Method: Non-Probability Sample
Enrollment: 657 (Actual)
Dates: Start 1998-10; Primary Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Change in cumulative daily doses of Sifrol® | up to 8 weeks
  Changes in the doses between visits are evaluated using Wilcoxon's signed rank test
Changes in cumulative daily doses of L-dopa | up to 8 weeks
  Changes in the doses between visits are evaluated using Wilcoxon's signed rank test

SECONDARY OUTCOMES:
Change from Baseline in Short Parkinson Evaluation Scale (SPES) total score | Baseline, after 8 weeks
Change from Baseline in SPES subscales | Baseline, after 8 weeks
  Psychopathological disturbances, Activities of daily living, Evaluation of motor function, Tremor, Resting Tremor, Postural tremor, Complications of therapy
Change from Baseline in Snaith-Hamilton-Pleasure-Scale total score | Baseline, after 8 weeks
  patients with SPES depression >= 2
Change from Baseline in Tremor Impact Scale (TIS-D) total score | Baseline, after 8 weeks
Change from Baseline in global Parkinson's Disease (PD) symptoms | Baseline, after 8 weeks
  Akinesia, anhedonia, depression, dyskinesia, motor fluctuation, cognitive disturbances, rigor and tremor
Global assessment of efficacy by investigator on a 5-point scale | after 8 weeks
Global assessment of tolerability by investigator on a 5-point scale | after 8 weeks
Number of patients with adverse events | up to 8 weeks
Number of patients with adverse drug reactions | up to 8 weeks